CLINICAL TRIAL: NCT03565614
Title: Reablement Intervention for Older Adults Conducted by a Multi Professional Home Rehabilitation Team: A Randomized Controlled Trial (RCT) With Qualitative Follow-ups of the Intervention
Brief Title: Reablement Intervention for Older Adults Conducted by a Multi Professional Home Rehabilitation Team
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mälardalen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IHR (Reablement)
Record Dates: First submitted 2017-12-18; First posted 2018-06-21 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Rehabilitation by Recovery of Function
Keywords: reablement; older people; personal care services; rehabilitation; multimorbidity; disability

STUDY DESIGN:
Intervention Model Description: Older adults (65+) applying for social care and services delivered by a municipality (Eskilstuna) in the county of Södermanland, Sweden. Presumptive participants are identified by the municipality care mangers. After informed consent, the users are randomized to either the intervention or control group. Exclusion criteria: Life-threatening disease, diagnosed mental illness, or severe cognitive dysfunction that would prevent the participant from expressing wants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reablement rehabilitation (Experimental): Reablement rehabilitation to maintain or increase the participants' physical, psychological and social functional abilities.
  Interventions: Behavioral: Reablement
- Traditional home care (Active Comparator): The traditional home care and required rehabilitation efforts as by the municipality's current practice.
  Interventions: Behavioral: Traditional home care

INTERVENTIONS:
Behavioral: Reablement — Intensive home-based rehabilitation is delivered up to 3 months by an interprofessional team (nurse, enrolled nurse, physiotherapist, occupational therapist, social worker). The entire team completed a 5-week college course. The team negotiates goal-directed contents of the rehabilitation initiatives with the user. Each user is handled deliberately based on decisions in the team in cooperation with the care managers overarching goals in admitted services. All participants have personal contact persons, and these contact persons have twice the time per participant as compared to traditional home care. The interprofessional team also has regular meetings to discuss every participant, and all rehabilitation goals activities related to those are documented.
  Arms: Reablement rehabilitation
Behavioral: Traditional home care — Traditional home care and required rehabilitation efforts as by the municipality's current practice. Includes the same professions as is included in the reablement intervention, but the team has had no joint college course, does not use the systematic goal-directed and negotiated approach as the reablement intervention, and has about half the time per participant as compared to the reablement intervention.
  Arms: Traditional home care

SUMMARY:
Background: People live increasingly longer and are expected to function independently in their own homes to a greater extent than before. This puts great demands on the support given to older persons living at home, to be efficient and provide good conditions for them to manage on their own and experience good health. Short time goal directed reablement delivered by a multidisciplinary team is expected to strengthen the functional capacity and quality of life, while home care-hours and thus municipal expenditures decline. Theoretical focus of this project is related to international classification of functionality and disability (ICF) in which participation are understood as engagement in life situations and related to the environment as well as the person. Reablement is expected to extend the time of independent and autonomous life for older persons while also reducing municipal costs of elder care.

Aim: This research project measures the effects of reablement in terms of bio-psycho-social health among older people (65+). In addition, the project highlights older person's experiences of the intervention and the professional team´s experiences of working with reablement.

Methods: This is a randomized controlled study of the intervention reablement performed by the multiprofessional team with controls receiving usual home care. The effects are measured by self-reported health and quality of life, physical capacity, and home care hours. Data are collected at inclusion (applying for home care), after the three months intervention and at six months. Interviews with users are performed after the intervention, and staff experiences through written narratives.

Impact of results: This project will contribute with collecting possible evidence of reablement, and contribute with knowledge development of older persons' bio-psycho-social health and experiences.

ELIGIBILITY:
Inclusion Criteria:

* older adults, over 65 years
* residing in the central areas of Eskilstuna municipality
* applying for social care and services delivered by the municipality of Eskilstuna

Exclusion Criteria:

* life-threatening disease
* severe mental illness
* severe cognitive dysfunction
* other conditions that prevent the participants from expressing their will or desires

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Change in self-assessed overall life satisfaction | Change from baseline overall life satisfaction rating at 6 months
  Participants' overall life satisfaction ratings are included in the Health as Ability of Acting questionnaire (HACT; Snellman et al. 2011), which is based on Nordenfelt's theory of health (2004). These global ratings are made on a VAS scale, which is coded from 0 (very unsatisfied with life) to 100 (very satisfied with life).

SECONDARY OUTCOMES:
Change in self-assessed general health | Change from baseline self-assessed general health ratings at 6 months
  Self-assessed general health is measured with an overall rating from the EQ-5D-5L (Herdman et al., 2011). These global ratings are made on a VAS scale, which is coded from 0 (the best health you can imagine) to 100 (the worst health you can imagine).
Change in self-assessed health-related quality of life | Change from baseline health-related quality of life ratings at 6 months
  Self-assessed health-related quality of life in five dimensions, i.e. mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, is measured with EQ-5D-5L (Herdman et al., 2011). Each of the five dimensions is rated on a five level response scale, which is coded and reported from 1 (no problems) to 5 (extreme problems).
Change in self-assessed mental health | Change from baseline mental health ratings at 6 months
  Mental health is mirrored with a short version of the Clinical Outcomes in Routine Evaluation - Outcome Measure (CORE-OM; Elfström et al. 2013, Evans, et al., 2002), called General Practitioner (GP-)CORE (Sinclair et al. 2005). The 14 items in GP-CORE are summarized and divided by 14, forming a total mean score ranging from 0 (no psychological distress) to 4 (maximum psychological distress).
Change in self-assessed health with respect to personal priorities | Change from baseline self-assessed health with respect to personal priorities at 6 months
  Participants' ratings from the Health as Ability of Acting questionnaire (HACT; Snellman et al. 2011) are categorized into one of three health groups:
  Good health: (a) Fulfilled vital goals or (b) the person possesses the ability to achieve the unfulfilled vital goals and the intention to use this ability or (c) experiencing a certain degree of ability to achieve vital goals and have the intention to use the ability.
  Acceptable health: (a) Unfulfilled vital goals. The person have a certain degree of ability to achieve goals and the intention to use the ability. (b) Unfulfilled vital goals. The person have a certain degree of ability to achieve these goals but have no intention to use the ability.
  Poor health: (a) experiencing a certain degree of ability to achieve vital goals, judged as important, and the intention to use the ability. (b) Unfulfilled vital goals. The person lacks the ability to achieve the unfulfilled goal or goals, despite judging them as important.
Change in self-assessed activity performance satisfaction | Change from baseline activity performance satisfaction ratings at 6 months
  Self-assessed activity performance satisfaction is estimated with interviewer administered Canadian Occupational Performance Measure (COPM; Law et al., 1990). In relation to a central activity problem area that the participants' themselves chose during the interview, the participants' are asked how well they think they can perform up to the five most important activities that relate to the central activity problem area. Then the participants are asked how satisfied they are with their performance, rating each activity performance satisfaction from 1 to 10. Then a mean value is calculated by dividing the sum of activity performance satisfaction ratings by the number of rated activities, giving a mean that can range from 1 (not at all satisfied) to 10 (extremely satisfied).
Change in self-assessed activity performance | Change from baseline activity performance ratings at 6 months
  Self-assessed activity performance is estimated with interviewer administered Canadian Occupational Performance Measure (COPM; Law et al., 1990). In relation to a central activity problem area that the participants' themselves chose during the interview, the participants' are asked how well they think they can perform up to the five most important activities that relate to the central activity problem area. The participants rate each activity from 1 to 10 regarding how well the can perform the activity. Then a mean value is calculated by dividing the sum of activity performance by the number of activities, giving a mean that can range from 1 (cannot perform the activity at all) to 10 (can perform the activity extremely well).
Change in lower extremities physical activity performance | Change from baseline lower extremities physical activity performance at 6 months
  Lower extremities physical activity performance is measured by a trained administrator with the Short Physical Performance Battery (SPPB; Guralnik et al., 1994). The SPPB is calculated from three components: the ability to stand for up to 10 seconds with feet positioned in three ways; time to complete a 3-m walk; and time to rise from a chair five times. Each component is scored from 0 to 4, with the scores from the three tests summed to give a total, with a maximum of 12 and a minimum of 0. A higher score indicates a higher level of function, while lower scores indicate a lower level of function.
Change in upper extremities physical activity performance | Change from baseline upper extremities physical activity ability at 6 months
  Upper extremities physical activity performance is measured with a hand dynamometer test (Mathiowetz et al., 1985). The Jamar hydrolic hand dynamometer model J00105 is used. The test of each hand is repeated 3 times, and the average is scored by the trained administrator as the recorded result. The resulting grip strength may vary from 0 kilograms (no grip strength) to 90 kilograms (maximum grip strength).

OTHER OUTCOMES:
Number of home care hours needed at 6 months | Home care hours needed at 6 months
  The number of home care hours needed is collected through the municipality's database. The number may vary from 0 hours (no home care needed) to 300 hours (in need of housing with personnel round the clock).

CONTACTS AND LOCATIONS:
Overall Officials: Lena-Karin Gustafsson, PhD, Principal Investigator — Mälardalen University
Locations (1):
- Eskilstuna municipality, Care and social care service, Rehabilitation unit, Eskilstuna, Södermanland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The unidentified research material will be available for 10 years after the research results have been publicized and then destroyed.
Access Criteria: If other researchers or authorities request access to the research material for review, Mälardalen University will examine the disclosure with accuracy. For example, the Privacy Act (2009: 40) will allow confidentiality of sensitive data is taken into account.

REFERENCES:
- [Derived] Gustafsson LK, Soderman M, Johansson C, Elfstrom ML. Interprofessional homebased reablement intervention for older adults in Sweden: a randomized controlled trial. BMC Geriatr. 2025 Apr 10;25(1):242. doi: 10.1186/s12877-025-05886-w. PMID 40211212